CLINICAL TRIAL: NCT06743204
Title: The Integrated Female Sexually Transmitted Infection Testing for HIV Epidemic Control Through PrEP (IN-STEP) Study
Acronym: IN-STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Abbott (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00447136; R01AI177132 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Gonorrhea Female; Chlamydia Females; Syphilis Female; Trichomonas Vaginalis; HIV; PrEP Uptake
Keywords: Sexually Transmitted Infections (STI); Diagnostics; HIV; Women; Africa; Uganda; PrEP; Adolescent Girls and Young Women (AGYW)
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-STEP Intervention (Experimental)
  Interventions: Other: Self-Reported Risk Screening for PrEP and Diagnostic STI testing
- Standard-of-Care (Active Comparator)
  Interventions: Other: Self-reported risk screening for PrEP and syndromic management for STIs

INTERVENTIONS:
Other: Self-Reported Risk Screening for PrEP and Diagnostic STI testing — The intervention arm will include: 1) Standard-of-care STI symptom screening: The investigators will ask participants if any STI symptoms 2) PrEP screening (if HIV- only): PrEP eligibility screening will be done using the standard-care Ministry Health self-reported risk screening (SRST) tool for PrEP 3) STI laboratory diagnostic testing: Regardless of HIV serostatus, vaginal swabs will be collected to test for chlamydia, gonorrhea, trichomonas, and human papilloma virus. Syphilis testing will be performed using blood samples participants provided in the Rakai Community Cohort Study. Participants who test positive for a curable sexually transmitted infection (chlamydia, gonorrhea, trichomonas, or syphilis) OR who screen eligible for PrEP using the Ministry of Health SRST AND are HIV- will be referred for same-day PrEP initiation. Participants who have symptoms indicative of STIs or who test positive for an STI will be provided with free treatment, as will the partner(s).
  Arms: IN-STEP Intervention
Other: Self-reported risk screening for PrEP and syndromic management for STIs — This active comparator (control) arm will receive the following: 1) Standard-of-care STI symptom screening: Regardless of HIV serostatus, participants will be asked if any STI symptoms 2) Syphilis testing for pregnant participants: Regardless of HIV serostatus, syphilis testing will be performed using blood samples provided in the Rakai Community Cohort Study. 3) PrEP screening (if HIV- only): Participants will be screened for PrEP eligibility using the standard-care Ministry Health self-reported risk screening (SRST) tool for PrEP. Participants who screen eligible for PrEP using the Ministry of Health SRST OR pregnant participant's who test positive for syphilis AND are HIV- will be referred for same-day PrEP initiation. Participants who have symptoms indicative of STIs or who test positive for syphilis will be provided with free treatment, as will the partner(s).
  Arms: Standard-of-Care

SUMMARY:
Globally, new HIV infections are concentrated in eastern and southern Africa where the infections are largely acquired by women outside of known key populations. Identifying African women at high risk for HIV acquisition and successfully engaging them in HIV prevention services, particularly pre-exposure prophylaxis (PrEP) programs, is an urgent global health priority. The U.S. President's Emergency Plan for AIDS Relief program in Africa typically relies on self-reported risk screening tools (SRST) to target HIV testing and refer individuals for PrEP. However, these tools have low to moderate sensitivity, missing many women at high risk for HIV. This is partly due to underreporting of risk factors, but also because many African women are at heightened HIV risk solely through relationships with high-risk male partners. Moreover, many African women enrolled into PrEP programs stop using PrEP within months of initiation. Decades of research shows that curable sexually transmitted infections (cSTI) are objective markers of future HIV risk, but cSTI testing largely has been omitted from African HIV programs. With the advent of lower cost multiplex cSTI testing and point of care diagnostics, there is new opportunity to determine whether integrating female cSTI testing services into HIV programs can improve HIV epidemic control. Here, the investigators will conduct an individually randomized effectiveness implementation trial of SRST plus cSTI diagnostic testing for chlamydia, gonorrhea, trichomonas, and syphilis compared to SRST alone to increase PrEP use among cis-gender African women aged 15-39 years. The investigators hypothesize that cSTI testing will increase PrEP use primarily through (i) improved identification of women at high risk for HIV and (ii) enhancement of self-perceived HIV risk. The proposed research will be nested within the Rakai Community Cohort Study, a population-based HIV surveillance cohort in Uganda. In Aim 1, ~4,500 HIV-negative women will be individually randomized 1:1 to PrEP screening based on SRST plus cSTI diagnostic testing (intervention) versus PrEP screening based on SRST alone (control arm). Both arms will be offered syndromic case management for cSTIs and syphilis testing for pregnant women (standard of care). The primary outcomes will be PrEP uptake, adherence, and persistence, assessed through clinical records and drug level testing. In Aim 2, the investigators will perform a mixed-methods, implementation science evaluation of female cSTI testing for HIV prevention and control. The investigators will use qualitative and quantitative methods to assess the mechanisms, barriers, and facilitators to improving PrEP outcomes through cSTI testing and how this varies by cSTI pathogen, SRST outcomes, and demographic profiles. In Aim 3, the investigators will use mathematical models to evaluate different cSTI testing approaches to reduce HIV incidence at a population level by considering what cSTIs to screen for, in what health care settings, and at what cost thresholds. The investigators will also model broader health benefits of cSTI testing. Results from this study will provide actionable, population-level information to inform strategic delivery of high impact HIV prevention through integrated HIV and cSTI programming in Africa.

DETAILED DESCRIPTION:
Globally, new HIV infections are concentrated in eastern and southern Africa and are largely acquired by women outside of known key populations. Identifying African women at highest risk for HIV acquisition and successfully engaging them in HIV prevention services, particularly pre-exposure prophylaxis (PrEP) programs, is an urgent global health priority. The U.S. President's Emergency Plan for AIDS Relief (PEPFAR) programs in Africa typically rely on self-reported risk screening tools (SRST) to target HIV testing and refer individuals for PrEP. However, these tools often perform poorly in validation studies, missing many women at high-risk for HIV acquisition. This is partly due to underreporting of risk factors, but also because many African women are at heightened HIV risk solely through monogamous relationships with high-risk male partners (i.e., network-based risk). Moreover, even among those African women referred and enrolled into PrEP programs, the vast majority stop using PrEP within several months of initiation. While PrEP discontinuation has been linked to various factors, lack of self-perceived HIV risk has been identified as a major barrier to PrEP use among cis-gender African women.

Here, the investigators hypothesize that compared to SRST alone, SRST integrated with diagnostic testing for curable sexually transmitted infections (cSTI) will increase PrEP use (uptake, adherence, and persistence) among cis-gender African women. The investigators further hypothesize that this increased PrEP use will occur through two primary mechanisms: (1) improved identification of women at high risk for HIV via objective biomarker screening, and (2) enhanced self-perceived HIV susceptibility among women with cSTIs. Decades of research has shown strong and consistent links between cSTIs and female HIV acquisition risk, but cSTI testing and treatment has been largely omitted from African HIV programs, partly due to lack of affordable cSTI diagnostics and laboratory capacity. In addition to being risk factors for HIV acquisition, cSTIs are also a significant cause of female reproductive morbidity, still birth, and neonatal morbidity and mortality. With the advent of lower cost multiplex cSTI testing and point of care diagnostics, there is new opportunity to determine whether integrated female cSTI testing can improve HIV epidemic control.

To test the central hypothesis, the investigators will conduct an individually randomized effectiveness implementation trial of SRST plus cSTI diagnostic testing for chlamydia, gonorrhea, trichomonas, and syphilis compared to SRST alone to increase PrEP use among cis-gender African women aged 15 to 39 years. The investigators preliminary observational data suggest that there is a high burden of undiagnosed cSTIs among African women at high risk for HIV and that adding cSTI diagnostic testing to existing PrEP eligibility screening efforts would nearly double the number of PrEP eligible women. Preliminary data also show women with cSTI symptoms are more likely to perceive themselves as being at high HIV risk, and that women diagnosed with cSTIs are more likely to use PrEP. The trial will be nested within the Rakai Community Cohort Study (RCCS), a population-based HIV surveillance cohort in the Lake Victoria basin of Uganda in Eastern Africa, a region with among the highest female HIV case burdens worldwide. Using a population-based design, the investigators will be able to determine what groups and in what programmatic settings cSTI testing would yield the greatest benefit for HIV epidemic control and overall population health. Specific aims are:

1. To conduct an individually randomized effectiveness implementation trial of SRST plus cSTI testing to increase PrEP use among African women at high HIV risk. ~4,500 HIV-negative women will be randomized 1:1 to PrEP eligibility screening based on SRST plus cSTI testing (intervention) versus screening based on SRST alone (control arm). Primary outcomes will be PrEP uptake after screening and adherence and persistence at 6 months assessed through survey, clinical records, and drug level testing.
2. To perform a mixed-methods, implementation science evaluation of female cSTI testing for improving PrEP use for HIV prevention. Guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, the investigators will use qualitative and quantitative methods to assess the mechanisms, barriers, and facilitators to improving PrEP outcomes through cSTI testing and how this varies by cSTI pathogen, SRST outcomes, and demographic profiles. Implementation science-focused modules will be added to the RCCS. In-depth qualitative interviews will be conducted at 1 and 6 months on a sample of participants after screening in both study arms.
3. To determine the most efficient, population-level female cSTI testing strategies to reduce HIV incidence in African settings. The investigators will use data and results from Aims 1 and 2 to inform mathematical models which will evaluate different cSTI testing approaches to reduce HIV incidence at a population level by considering what cSTIs to screen for, in what health care settings, and at what cost thresholds.

IMPACT: The proposed research will provide a novel and rigorous understanding of whether integrated cSTI diagnostic testing can facilitate female PrEP use in order to reduce HIV incidence through the identification of underserved women at high risk for HIV acquisition and enhancement of their self-perceived HIV susceptibility. Study results will provide actionable, Randomized Controlled Trial (RCT) level, and population-level information to inform strategic delivery of high impact HIV prevention interventions through integrated HIV and cSTI programming.

ELIGIBILITY:
Inclusion criteria:

* Sexually active females aged 15-39 years,
* resident in Rakai Community Cohort Study (RCCS) communities and who have participated in the most recent RCCS survey will be eligible to participate irrespective of their HIV serostatus.
* Pregnant women will be included in this study
* Additionally, eligibility criteria include participation in the most recent RCCS with consent to store and test plasma specimens collected during the RCCS visit,
* consent to be re-contacted for future studies, and
* willingness to be randomized in IN-STEP.

Exclusion criteria:

* Individuals incapable of providing consent or
* not meeting the above criteria will be excluded from the study.

Ages: 15 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5560 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
PreP uptake | From enrollment up to 3 months post enrollment
  PrEP uptake will be defined as the proportion of HIV-negative women initially not taking PrEP at baseline who initiated PrEP by 3 months as determined from IN-STEP survey and clinical records.
PreP adherence | From enrollment up to 6 months post enrollment
  PrEP adherence will be defined as the proportion of HIV-negative women initially not taking PrEP with high-level adherence. Tenofovir diphosphate (TFV-DP) ≥800 fmol/punch at the 6-month IN-STEP visit.
PreP persistence | From enrollment up to 6 months post enrollment
  PrEP persistence will be defined as the proportion of HIV-negative women initially not taking PrEP with continuous attendance at quarterly PrEP program follow-up/refill visits through 6 months after PrEP initiation as validated through clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kathryn Grabowski, Associate Professor, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The Rakai Health Sciences Program (RHSP) has a written policy on the sharing of data and of laboratory specimens. Institutions, groups or researchers who propose to use Rakai data or specimens are required to submit a brief proposal/data request form describing the goals and methods of the proposed analyses. Based on this document and additional discussions with the party(ies) proposing the collaboration, the decision as to whether and/or how to proceed is made by consensus between senior Ugandan and US-based Investigators. The decision takes into account Uganda Ministry of Health directives regarding the maximization of research findings and safeguards regarding misuse, misappropriation or misinterpretation of data. Feasibility, availability of resources (such as Rakai Program analysts' time to help prepare and anonymize data sets to ensure no potential loss of confidentiality), and research importance/priority are also taken into consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of study outcomes
Access Criteria: E-mail PI